CLINICAL TRIAL: NCT04481373
Title: Targeting HIV Retention and Improved Viral Load Through Engagement ('THRIVE')
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: University of Iowa (Other); Brown University (Other); University of Texas (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Thomas Giordano, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-47444; 5R34MH122294 (NIH)
Record Dates: First submitted 2020-07-09; First posted 2020-07-22 (Actual); Results first posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Human Immunodeficiency Virus; Depression; Anxiety
Keywords: Acceptance and Commitment Therapy; HIV; depression; anxiety; distress; avoidance
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Depression; Anxiety Disorders | interventions — Nicotine; Educational Status; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- THRIVE (Experimental): Acceptance and Commitment Therapy plus Education about HIV A master's level mental health professional will provide the 4-5 hour intervention for out-of-care PWH during a hospitalization. There are two important components to the intervention: Acceptance and Commitment Therapy (ACT) content, targeting avoidance with acceptance-based coping and active engagement in values-based living, and HIV education.
  Interventions: Behavioral: THRIVE
- Treatment as Usual (Other): Patients get usual care at the hospital. Service linkage workers (SLWs) meet with all hospitalized PWH and cover educational aspects of the care.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: THRIVE — The ACT components (3-3.5 hours) will focus on clarifying patient values and goals and identifying obstacles that may be getting in the way of living a rich life. Short-and long-term effects of avoidance will be discussed (e.g., avoidance reduces immediate contact with distressing experiences and provides short-term relief but leads to greater dysfunction in long run). Patients will be taught acceptance, mindfulness, and perspective taking to help patient cope with difficult emotions and thoughts that may interfere with living a values-driven life. Individuals will also be encouraged to examine the costs of stigmatization on their life (e.g. avoidance of medical care, sense of isolation).
  Education will include medical information about HIV, services available at the clinic, and health needs related to comorbidities. This content to be delivered in 30 minutes.
  Other Names: Acceptance and Commitment Therapy plus Education
  Arms: THRIVE
Other: Treatment as Usual — Patients get usual care at the hospital. Service linkage workers (SLWs) meet with all hospitalized PWH and cover educational aspects of the care.
  Arms: Treatment as Usual

SUMMARY:
Many people with HIV infection are not consistently engaged in outpatient HIV care, and avoidance, stigma and denial contribute to poor engagement in HIV care. This project will develop and pilot test a new intervention, "THRIVE," for hospitalized persons who are out of HIV care and endorse avoidance, to improve how well they stay in outpatient HIV care after discharge. If successfully developed, the intervention will undergo large scale testing in later studies and could improve the health of persons with HIV infection and help end the HIV epidemic in the United States.

DETAILED DESCRIPTION:
Poor retention in HIV primary care results in lower rates of HIV viral suppression, higher rates of HIV transmission, and exacerbates racial and ethnic disparities in health outcomes, including survival. To date, there are no interventions that effectively relink and retain PWH in care when they are found outside the HIV clinic. Many persons with HIV infection (PWH) are hospitalized with life-threatening but preventable complications of inadequately treated HIV infection. They are among the most important patients to retain in care. Our previous research shows that among PWH who are out of care and hospitalized, avoidance coping, stigma, and mental health difficulties were nearly universal. Further, avoidance coping was a predictor of failure to re-engage in care after discharge. Acceptance and Commitment Therapy (ACT) is a transdiagnostic intervention with the capacity to address a range of psychosocial and behavior-related issues that PWH experience. ACT helps patients overcome avoidance, particularly avoidance of uncomfortable internal states and the situations that trigger such states, by promoting acceptance-based coping and re-engagement in meaningful and valued-life activities. Brief ACT interventions appear to be feasible, acceptable, and at least preliminarily, have efficacy. The investigators propose to develop, refine, and pilot a brief (4-5 contact hours) ACT intervention for hospitalized, out-of-care PWH. 'Targeting HIV Retention and Improved Viral load through Engagement' ('THRIVE') will aim to help patients overcome avoidance, a maladaptive coping strategy implicated in a range of problems, including depression, anxiety, substance abuse, and HIV-related self-stigma, all of which constitute barriers to care. Delivering THRIVE in the hospital with a phone booster session after discharge will increase therapy initiation and completion, the lack of which is often the greatest obstacle to effective delivery of mental health services for PWH. In Aim 1, a brief hospital-based transdiagnostic, individually delivered ACT intervention (THRIVE) tailored specifically for out-of-care hospitalized PWH will be developed. Input from a multi-disciplinary team of expert care providers and PHW will be utilized to create the therapist protocol and patient workbook. The investigators will then pilot THRIVE in 10 hospitalized out-of-care PWH who will provide qualitative feedback on the intervention. The feedback, along with input from patients and the multi-disciplinary team, will be used to refine THRIVE. In Aim 2, the investigators will conduct a pilot randomized clinical trial (RCT) of the refined THRIVE intervention (N=35) compared to treatment as usual (N=35). This pilot RCT will 1) evaluate feasibility and acceptability for a full-scale RCT; and 2) examine trends in outcomes of interest for the definitive RCT. The investigators will then be positioned to submit a separate grant to test the efficacy of THRIVE in a fully powered randomized trial. This work has the potential to decrease HIV morbidity and racial/ethnic disparities and contribute to ending the HIV epidemic in the United States, which are NIH priorities.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized at Ben Taub Hospital, Houston, TX;
* at least 18 years of age;
* able to speak English or Spanish;
* HIV infected;
* able to provide informed consent and participate in the study (patients who are temporarily unable to participate will be followed and approached for enrollment if and when they are cognitively and physically capable of consenting and participating);
* HIV VL>1000 c/mL;
* never in care or currently out of HIV care, defined as not meeting the 'visit constancy' measure (≥1 completed HIV primary care visit at Thomas Street Health Center (TSHC), Houston, TX, in each of the three 4-month intervals preceding admission); or ≥2 "no shows" to HIV primary care visits at TSHC in the last year.
* endorse one of two avoidance coping statements with the highest factor loadings on the Avoidant Coping Subscale from the Coping with HIV/AIDS scale

Exclusion Criteria:

* intending to use a source of HIV primary care other than TSHC after discharge, because their outcomes cannot be evaluated;
* in the opinion of the primary medical team caring for the patient, likely to be discharged to an institutional setting, die in the hospital or enter hospice;
* incarcerated or expected to be discharged to prison or jail;
* enrolled in another research study with prospective follow-up;
* pregnant, since pregnant women receive additional efforts to be linked and retained in care;
* admitted with acute psychosis which would preclude informed consent or meaningful participation with the intervention.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lilian Dindo, Ph.D, Principal Investigator — Baylor College of Medicine; Thomas Giordano, M.D., M.P.H., Principal Investigator — Baylor College of Medicine
Locations (1):
- Ben Taub Hospital, Houston, Texas, United States

REFERENCES:
- [Background] Dindo L, Moitra E, Roddy MK, Ratcliff C, Markham C, Giordano T. Development and Initial Feasibility of a Hospital-Based Acceptance and Commitment Therapy Intervention to Improve Retention in Care for Out-of-Care Persons with HIV: Lessons Learned from an Open Pilot Trial. J Clin Med. 2022 May 17;11(10):2827. doi: 10.3390/jcm11102827. PMID 35628955

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | THRIVE | Treatment as Usual
Started | 39 | 36
Completed | 35 | 35
Not Completed | 4 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Viral load in hospital not over 1000 | 2 | 1
Not completed — Death before hospital discharge | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | THRIVE | Treatment as Usual | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.2 (12.3) | 42.1 (11.8) | 44.7 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 27 | 28 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 18 | 20 | 38
  White | 15 | 13 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 9 | 18
  Not Hispanic or Latino | 26 | 26 | 52
  Unknown or Not Reported | 0 | 0 | 0
Coping with HIV/AIDS Scale - Positive Coping [Median (Inter-Quartile Range); unit: units on a scale] — The coping with HIV/AIDS positive coping scale scores range between 0 and 5. There are 5 questions in the positive coping subscale. Each question answered "often or a lot of the time" counts as one point. A higher total sum suggests more positive coping, which is beneficial.
  units on a scale | 2 [1 to 4] | 3 [2 to 4] | 2 [2 to 4]
Coping with HIV/AIDS Scale - Avoidance Coping [Median (Inter-Quartile Range); unit: units on a scale] — The coping with HIV/AIDS avoidance coping scale scores range between 0 and 9. There are 9 questions in the avoidance coping subscale. Each question answered "often or a lot of the time" counts as one point. A higher total sum suggests more avoidance coping, which is not beneficial.
  units on a scale | 2 [1 to 4] | 3 [2 to 5] | 3 [2 to 5]
Coping with HIV/AIDS Scale - Seeking Social Support Subscale [Count of Participants; unit: Participants] — There are 2 questions in the seeking social support subscale. We report the number of participants who answer each question "often or a lot of the time". More responses "often or a lot of the time" suggests seeking more social support, which is beneficial.
  Participants
    Seeking Social Support - "Often" or "a lot" for 1 of the 2 subscale items | 10 | 6 | 16
    Seeking Social Support - "Often" or "a lot" for 2 of the 2 subscale items | 1 | 3 | 4
Internalized AIDS-Related Stigma Scale (IARSS) [Median (Inter-Quartile Range); unit: units on a scale] — The Internalized AIDS-Related Stigma Scale (IARSS) is a 6-item scale with scores that range between 0 and 6. There are 6 questions in the stigma scale. Each question answered "yes" counts as one point. A higher total sum suggests more internalized stigma, which is not beneficial.
  units on a scale | 2 [1 to 4] | 3 [2 to 5] | 3 [2 to 4]
Depression Anxiety and Stress Scale (DASS-21) [Median (Inter-Quartile Range); unit: units on a scale] — The Depression Anxiety and Stress Scale (DASS-21) has 21 items. Each item is scored 1, 2, or 3. The score is calculated by adding each item's score, multiplied by 2. The range of scores for the total scale is between 0 and 126. Each subscale (depression, anxiety, and stress) has 7 items with a range of scores between 0 and 42. Higher scores suggest higher depression, anxiety, and stress, which are not beneficial.
  units on a scale
    DASS-21 Depression | 8 [6 to 16] | 10 [2 to 18] | 10 [4 to 16]
    DASS-21 Stress | 10 [4 to 18] | 10 [2 to 16] | 10 [4 to 18]
    DASS-21 Anxiety | 10 [4 to 14] | 10 [4 to 18] | 10 [4 to 16]
    DASS Total | 26 [20 to 48] | 36 [14 to 48] | 31 [18 to 48]
AUDIT (Hazardous Alcohol Use) [Count of Participants; unit: Participants]
  Alcohol use (at least monthly) | 20 | 10 | 30
  Consumption at Hazardous level | 7 | 6 | 13
Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) [Count of Participants; unit: Participants]
  Ever Used Tobacco products | 19 | 23 | 42
  Ever Used Alcoholic beverages | 29 | 27 | 56
  Ever Used Cannabis/Cocaine/Amphetamine/Inhalants/S | 35 | 33 | 68
  Used in past 3 months Tobacco products | 14 | 10 | 24
  Used in past 3 months Alcoholic beverages | 7 | 2 | 9
  Used in past 3 months Cannabis/Cocaine/Amphetamine | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Enrollment and Randomization: Eligible But Declined Participation
Description: The number of eligible PWH who agree and decline to participate, and reasons for declining;
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | THRIVE | Treatment as Usual
Number analyzed (Participants) | 39 | 36
Participants | 0 | 0

2. Primary Outcome: Acceptability of Enrollment and Randomization: Completion Sessions
Description: Completion of at least 3 out of 4 intervention sessions in the THRIVE group
Time Frame: 6 months
Population: 80% of THRIVE participants received at least 3 of 4 sessions. Participants randomized to the Treatment as Usual arm were not analyzed and did not receive the intervention (sessions).
Measure: Count of Participants; unit: Participants
Groups:
- Treatment as Usual: Patients get usual care at the hospital. Service linkage workers (SLWs) meet with all hospitalized PWH and cover educational aspects of the care. Participants randomized to the Treatment as Usual arm were not analyzed and did not receive the intervention (sessions).
Arm/Group | THRIVE | Treatment as Usual
Number analyzed (Participants) | 35 | 0
Participants | 28 | 0

3. Primary Outcome: Acceptability of the Intervention: 6 Month Follow-up
Description: The completion of participant 6-month follow-up assessments
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | THRIVE | Treatment as Usual
Number analyzed (Participants) | 35 | 35
Participants | 21 | 26

4. Primary Outcome: Acceptability of the Intervention
Description: Mean duration of contact for participants who completed all four sessions
Time Frame: 6 months
Population: Treatment as usual participants did not get any intervention.
Measure: Number; unit: minutes
Arm/Group | THRIVE | Treatment as Usual
Number analyzed (Participants) | 25 | 0
minutes | 135.5 |

5. Secondary Outcome: Viral Load Improvement
Description: Viral load less than 200 copies/mL at 180 days +/- 42 days of follow up
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | THRIVE | Treatment as Usual
Number analyzed (Participants) | 31 | 32
Participants | 12 | 14

6. Secondary Outcome: Number of Patients Who Are Retained in HIV Care
Description: Number of patients who complete at least 2 visits with an HIV clinician within 6 months, including 1 visit within 30 days of discharge
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | THRIVE | Treatment as Usual
Number analyzed (Participants) | 33 | 32
Participants | 13 | 16

7. Other Pre Specified Outcome: Internalized AIDS-Related Stigma Scale (IARSS)
Description: The Internalized AIDS-Related Stigma Scale (IARSS) is a 6-item scale with scores that range between 0 and 6. There are 6 questions in the stigma scale. Each question answered "yes" counts as one point. A higher total sum suggests more internalized stigma, which is not beneficial.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | THRIVE | Treatment as Usual
Number analyzed (Participants) | 21 | 26
units on a scale | 2 [2 to 5] | 3 [2 to 5]

8. Other Pre Specified Outcome: Depression Anxiety and Stress Scale (DASS-21).
Description: The Depression Anxiety and Stress Scale (DASS-21) has 21 items. Each item is scored 1, 2, or 3. The score is calculated by adding each item's score, multiplied by 2. The range of scores for the total scale is between 0 and 126. Each subscale (depression, anxiety, and stress) has 7 items with a range of scores between 0 and 42. Higher scores suggest higher depression, anxiety, and stress, which are not beneficial.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | THRIVE | Treatment as Usual
Number analyzed (Participants) | 21 | 26
units on a scale
  DASS-21 Total | 28 [16 to 48] | 32 [18 to 48]
  DASS-21 Depression | 8 [4 to 14] | 10 [2 to 18]
  DASS-21 Stress | 10 [6 to 16] | 12 [6 to 16]
  DASS-21 Anxiety | 8 [2 to 18] | 11 [8 to 16]

9. Other Pre Specified Outcome: Alcohol Use Disorders Identification Test (AUDIT)
Description: This 3-item screener that identifies problem alcohol use for both men and women. Participants respond on a 5-point scale. Higher numbers represent more difficulty.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | THRIVE | Treatment as Usual
Number analyzed (Participants) | 21 | 26
Participants
  Alcohol use (at least monthly) | 8 | 13
  Consumption at Hazardous level | 6 | 9

10. Other Pre Specified Outcome: The Alcohol, Smoking and Substance Involvement Screening Test (ASSIST)
Description: This measure asks about substance use of 7 categories of drugs in the previous 3 months and in a person's life time. Participants respond YES or NO to each category of drugs.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | THRIVE | Treatment as Usual
Number analyzed (Participants) | 21 | 26
Participants
  Ever Used Tobacco products | 10 | 13
  Ever Used Alcoholic beverages | 12 | 20
  Ever Used Cannabis/Cocaine/Amphetamine/Inhalants/Sedatives | 20 | 26
  Used in past 3 months Tobacco products | 7 | 11
  Used in past 3 months Alcoholic beverages | 4 | 3
  Used in past 3 months Cannabis/Cocaine/Amphetamine/Inhalants/Sedatives | 7 | 7

11. Other Pre Specified Outcome: Coping With HIV/AIDS Scale: Coping and Social Support
Description: The coping with HIV/AIDS positive coping scale scores range between 0 and 5. There are 5 questions in the positive coping subscale. Each question answered "often or a lot of the time" counts as one point. A higher total sum suggests more positive coping, which is beneficial.
  The coping with HIV/AIDS avoidance coping scale scores range between 0 and 9. There are 9 questions in the avoidance coping subscale. Each question answered "often or a lot of the time" counts as one point. A higher total sum suggests more avoidance coping, which is not beneficial.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: Medan, ICR
Arm/Group | THRIVE | Treatment as Usual
Number analyzed (Participants) | 21 | 26
Medan, ICR
  Coping with HIV - Positive Coping | 4 [3 to 4] | 3.5 [1 to 4]
  Coping with HIV - Avoidance Coping | 3 [1 to 5] | 3 [1 to 4]

12. Other Pre Specified Outcome: Coping With HIV/AIDS Scale
Description: There are 2 questions in the seeking social support subscale. We report the number of participants who answer each question "often or a lot of the time". More responses "often or a lot of the time" suggests seeking more social support, which is beneficial.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | THRIVE | Treatment as Usual
Number analyzed (Participants) | 21 | 26
Participants
  Seeking Social Support - Often/a lot for 1 of 2 items | 4 | 4
  Seeking Social Support - Often/a lot for 2 of 2 items | 2 | 2

13. Other Pre Specified Outcome: Client Satisfaction Questionnaire (CSQ)
Description: The Client Satisfaction Questionnaire (CSQ) scale has 8 items. Each item is scored 1, 2, 3, or 4. The score is calculated by adding each item's score. The range of scores for the total scale is between 8 and 32. Higher scores represent greater satisfaction with the THRIVE intervention.
Time Frame: 2 weeks
Population: CSQ was only measured in the THRIVE arm.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | THRIVE | Treatment as Usual
Number analyzed (Participants) | 27 | 0
units on a scale | 31 [26 to 31] |

ADVERSE EVENTS:
Time Frame: Enrollment through 6 months
Description: We are only reporting all-cause mortality, serious adverse events, and other adverse events attributable to the study assessments or intervention.
Arm/Group | THRIVE | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 2/35 | 1/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/73/NCT04481373/Prot_SAP_ICF_000.pdf